CLINICAL TRIAL: NCT06218342
Title: The Study of Henagliflozin in Relieving Progression of Type 2 Diabetes With Non-alcoholic Fatty Liver Disease
Brief Title: Henagliflozin in Relieving Type 2 Diabetes With Non-alcoholic Fatty Liver Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023412
Record Dates: First submitted 2023-11-21; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — henagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Henagliflozin (Experimental): Participants in this group will receive a combination of lifestyle intervention, background medication, and Henagliflozin. The choice of hypoglycemic drugs within the background medication is restricted to either one, two, or three among metformin, DPP-4 inhibitors, alpha-glucosidase inhibitors, or secretagogues.
  Interventions: Drug: Henagliflozin
- Control (Other): Participants in this group will receive lifestyle intervention and background medication. The choice of hypoglycemic drugs within the background medication is restricted to either one, two, or three among metformin, DPP-4 inhibitors, alpha-glucosidase inhibitors, or secretagogues.
  Interventions: Other: Background medication

INTERVENTIONS:
Drug: Henagliflozin — Besides lifestyle intervention and background medication, participants will be prescribed Henagliflozin at standard clinical doses.
  Arms: Henagliflozin
Other: Background medication — Participants will only receive lifestyle intervention and background medication.
  Arms: Control

SUMMARY:
This study is a randomized, non-blinded clinical trial specifically designed to assess the initial feasibility and efficacy of SGLT2 inhibitors in treating NAFLD among adults diagnosed with type 2 diabetes.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a metabolic liver disease that encompasses a spectrum of progressive pathological changes, ranging from simple steatosis to non-alcoholic steatohepatitis (NASH), cirrhosis, and hepatocellular carcinoma (HCC). Epidemiological data demonstrate a close association between type 2 diabetes and NAFLD. Approximately 49% to 62% of individuals with type 2 diabetes have concurrent NAFLD, and those with NAFLD have a risk of developing diabetes more than twice that of the general population. NAFLD not only increases the risk of developing type 2 diabetes but also accelerates the progression of diabetes-related target organ damage, leading to adverse metabolic and cardiovascular risks. Currently, there is a global lack of comprehensive public health strategies for addressing NAFLD, and clinically, there are still no approved drugs specifically for treating NAFLD.

NAFLD is diagnosed through abnormal liver function test results and imaging examinations. The NAFLD Fibrosis Score (NFS) and Fibrosis-4 (FIB-4) Index can be used for clinical screening of NASH in individuals with type 2 diabetes. Ultrasound attenuation parameters (UAP) and liver stiffness measurements (LSM) based on transient elastography (TE) can accurately differentiate between liver steatosis and the degree of liver fibrosis. This technique, known for its non-invasive, safe, and reproducible nature, has found widespread application in diagnosing the extent of liver fat and fibrosis in patients with chronic liver diseases.

The primary approach to treating NAFLD involves modifying poor lifestyle habits, however, lifestyle changes are often difficult to sustain in the long term. Currently, neither the U.S. FDA nor the European Medicines Agency has approved any medications specifically for NAFLD treatment. Given the central role of insulin resistance in the development of NAFLD, hypoglycemic medications have become a new focus in the prevention and treatment of NAFLD. Sodium-glucose co-transporter-2 (SGLT-2) inhibitors, by inhibiting SGLT-2 activity, reduce the reabsorption of glucose in the proximal renal tubules, causing excess glucose to be excreted in the urine, thereby lowering blood sugar. Reports suggest that SGLT-2 inhibitors also have several other beneficial effects, including reducing the risk of cardiovascular and kidney diseases, improving blood pressure control, aiding weight reduction, and lowering liver fat content. Previous studies have shown that SGLT-2 inhibitors can improve alanine transaminase, aspartate transaminase, gamma-glutamyl transferase, and the FIB-4 Index in patients with type 2 diabetes complicated by NAFLD, potentially exhibiting anti-fibrotic effects on the liver. Henagliflozin, the SGLT-2 inhibitor used in this study, is a compound independently developed with intellectual property by Jiangsu Hengrui Medicine Co., Ltd. Henagliflozin has demonstrated efficacy and safety in monotherapy for inadequately controlled type 2 diabetes patients with poor diet and exercise control or in combination with metformin for inadequately controlled type 2 diabetes patients.

This study aims to observe the clinical efficacy of henagliflozin treatment for type 2 diabetes complicated by NAFLD in individuals, evaluating its potential to improve liver fat changes and fibrosis indicators in NAFLD, promoting NASH regression, and alleviating the progression of liver fibrosis, building upon lifestyle changes and basic treatments. The secondary objectives include investigating the effects of henagliflozin on liver fat content, visceral fat area, liver enzymes, and blood sugar improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 70 years old.
* Diagnosed with type 2 diabetes according to World Health Organization (WHO) diagnostic criteria, with evidence of fatty liver on ultrasound, and FIB-4 index >1.3.
* Willing to participate in this study and sign an informed consent form. In case the subject lacks the ability to read the informed consent form (e.g., illiterate subjects), the informed process must be witnessed by a designated person who will sign the informed consent form.
* Have not used oral antidiabetic medications or have used one to three oral antidiabetic medications (limited to metformin, Dipeptidyl peptidase-4 (DPP-4) inhibitors, alpha-glucosidase inhibitors, or sulfonylureas) with an HbA1c between 7% and 10%, and fasting venous blood glucose ≤13.3 mmol/L.
* Have not used thiazolidinediones (TZDs), sodium-glucose co-transporter-2 inhibitors (SGLT-2i), glucagon-like peptide-1 receptor agonists (GLP-1RA), or other antidiabetic drugs that may affect liver fat content in the last 90 days.
* Weight change of less than 5% in the last 3 months.
* If of childbearing age, must use reliable contraceptive measures.

Exclusion Criteria:

* Daily alcohol intake of >30 g in the past 10 years or daily alcohol intake of >10 g in the last year.
* History of liver diseases such as hepatitis B, chronic hepatitis C, primary biliary cholangitis (PBC), biliary obstruction disorders, drug-induced liver damage, hemochromatosis, liver cirrhosis, autoimmune hepatitis.
* Patients with decompensated liver cirrhosis, concurrent liver cancer, HIV-positive status, or substance abuse.
* Type 1 diabetes.
* Participation in other clinical trials of diabetes treatment drugs in the 3 months prior to the start of this study.
* Occurrence of diabetic ketoacidosis, diabetic lactic acidosis, or hyperosmolar non-ketotic coma in the past 6 months.
* Occurrence of unexplained severe hypoglycemic events in the past 6 months (requiring assistance for recovery) or recurrent hypoglycemia: such as experiencing two or more low blood sugar events (blood glucose ≤3.9 mmol/L) in the month before screening.
* Severe heart disease patients, such as New York Heart Association (NYHA) class IV, unstable angina, or history of myocardial infarction.
* Abnormal liver function, with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 3 times the upper normal limit, or total bilirubin (TBIL) greater than 2 times the upper normal limit.
* Chronic kidney damage, with a creatinine level (Cr) >200 µmol/L or an estimated glomerular filtration rate (eGFR) <30 mL·min-1.
* Use of corticosteroid medications (excluding short-term topical or inhaled use).
* Patients with malignant tumors, active tuberculosis, or acute/chronic infections.
* Vulnerable populations, including pregnant women, individuals with mental illness, critically ill patients, individuals with cognitive impairments, etc.
* History of recurrent urinary tract infections or genital infections, or allergies to the investigational drug or its components.
* Patients assessed by the clinical doctor as having low blood volume.
* Patients deemed unsuitable for participation in this clinical study by the investigator, for reasons not covered above.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound attenuation parameter (UAP) | 24 weeks
  Changes in ultrasound attenuation parameter (UAP) from baseline. Higher UAP correlates with increased severity of steatosis.
Liver stiffness measurement (LSM) | 24 weeks
  Changes in liver stiffness measurement (LSM) from baseline. Higher LSM values correlate with advancement in the stage of liver fibrosis.

SECONDARY OUTCOMES:
Non-Alcoholic Fatty Liver Disease Fibrosis Score (NFS) | 24 weeks
  Changes in Non-Alcoholic Fatty Liver Disease Fibrosis Score (NFS) from baseline. Higher NFS score suggests advanced liver fibrosis.
Fibrosis Index Based on 4 Factors (FIB-4 Index) | 24 weeks
  Changes in FIB-4 Index from baseline. Higher FIB-4 Index correlates with increased severity of hepatic fibrosis.
Liver fat content | 24 weeks
  Changes in liver fat content from baseline
Liver enzymes | 24 weeks
  Changes in liver enzymes from baseline, the enzymes include ALP (alkaline phosphatase), ALT (alanine transaminase), AST (aspartate aminotransferase), and GGT (gamma-glutamyl transferase).
Cholestatic proteins (Chitinase 3-like protein 1, CHI3L1) | 24 weeks
  Changes in CHI3L1 from baseline. Higher CHI3L1 level suggests advanced liver fibrosis.
Intrabdominal fat | 24 weeks
  Changes in visceral fat area from baseline
Glucose level | 24 weeks
  Changes in HbA1c from baseline
Body weight | 24 weeks
  Changes in body weight from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqiang Zhou, Principal Investigator — Sir Run Run Shaw Hospital